CLINICAL TRIAL: NCT00002926
Title: Autologous Peripheral Blood Stem Cell Transplantation (PSCT) Versus a Second Intensive Consolidation Course After a Common Induction and Consolidation Course in Patients With Bad Prognosis Myelodysplastic Syndromes (MDS) and Acute Myelogenous Leukemia Secondary (SAML) to MDS of More Acute Than 6 Months Duration
Brief Title: Combination Chemotherapy With or Without Peripheral Stem Cell Transplantation in Treating Patients With Myelodysplastic Syndrome or Acute Myelogenous Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065336; EORTC-06961
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2001-05

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: secondary acute myeloid leukemia; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory cytopenia with multilineage dysplasia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Cytarabine; Etoposide; Idarubicin; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: cytarabine
Drug: etoposide
Drug: idarubicin
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of peripheral stem cell transplantation with high-dose cytarabine in treating patients with myelodysplastic syndrome or acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the value of autologous peripheral stem cell transplantation versus high dose cytarabine (Ara-C) performed after a common induction and consolidation course in patients with poor prognosis myelodysplastic syndromes (MDS) or acute myelogenous leukemia secondary to MDS.
* Compare the disease free survival and overall survival of patients who reached complete recovery according to the presence of an HLA-identical donor.
* Monitor cytogenetic and clonal remission after intensive antileukemic therapy including stem cell transplantation.
* Monitor residual disease and the hematopoietic clonal status of autologous peripheral blood stem cells mobilized after one consolidation course.
* Assess recovery time of granulocyte and platelet counts following each treatment step.

OUTLINE: Induction treatment with idarubicin on days 1,3,5; Ara-C from days 1 through 10; etoposide on days 1 through 5. On day 28 there will be assessment of responses. If there is at least partial response, the cycle will repeat the induction course for another 28 days. There is peripheral blood stem cell collection and cryopreservation following family HLA-typing. If there is no HLA match, then those who remained in remission after these consolidation courses will be randomized to either peripheral blood stem cell transplantation or HiDAC treatment.

PROJECTED ACCRUAL: 80 patients will be entered per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathological confirmation of one of the following:

  * Untreated refractory anemia with excess blasts (RAEB) in transformation
  * RAEB with greater than 10% blasts cells in the bone marrow
  * Other myelodysplastic syndromes
  * Profound cytopenias
  * Acute myelogenous leukemia (AML) supervening after overt myelodysplastic syndromes (MDS) of more than 6 months duration
* No blast crisis of chronic myeloid leukemia
* No leukemias supervening after other myeloproliferative disease
* No leukemias supervening after overt MDS of less than 6 months duration
* The following are allowed:

  * Secondary acute leukemias following Hodgkin's disease or other malignancies
  * Secondary leukemias following exposure to alkylating agents or radiation

PATIENT CHARACTERISTICS:

Age:

* 16-60

Performance status:

* WHO 0-2

Hematopoietic:

* If RAEB, blasts cells of greater than 10% in bone marrow
* Neutrophil count less than 5,000 or Platelet count less than 200,000
* Chronic myelomonocytic leukemia (CMML) with greater than 5% blasts cells in bone marrow, or CMML with neutrophil count greater than 160,000 or monocyte count greater than 2,600

Hepatic:

* Bilirubin no greater than 1.5 times normal

Renal:

* Creatinine no greater than 1.5 times normal

Cardiovascular:

* No patients with severe heart failure requiring diuretics or an ejection fraction of less than 50%

Neurological:

* No severe concomitant neurological disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No treatments within the past 4 weeks of:

  * Biological response modifiers AND/OR
  * Low dose Ara-C

Chemotherapy:

* No prior intensive treatment for MDS or AML

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior treatment for MDS or AML

Surgery:

* Not specified

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 1996-12

CONTACTS AND LOCATIONS:
Overall Officials: Theo De Witte, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (40):
- Belgium (8):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
- University Hospital Rebro, Zagreb, Croatia
- Institute of Hematology and Blood Transfusion, Prague, Czechia
- France (4):
  - Hopital Edouard Herriot, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hotel Dieu de Paris, Paris
  - Hopital Necker, Paris
- Germany (5):
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Medizinische Klinik und Poliklinik, Heidelberg
  - Klinikum Grosshadern, Munich (Muenchen)
  - Eberhard Karls Universitaet, Tübingen
- Ospedale San Eugenio, Rome, Italy
- Netherlands (10):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Medical Center Nijmegen, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Erasmus Medical Center, Rotterdam
  - Leyenburg Ziekenhuis, The Hague
  - Sophia Ziekehuis, Zwolle
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg (Goteborg)
  - University Hospital of Linkoping, Linköping
  - Orebro University Hospital, Örebro
  - Huddinge University Hospital, Stockholm
- Switzerland (6):
  - University Hospital, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen

REFERENCES:
- [Result] de Witte T, Hagemeijer A, Suciu S, Belhabri A, Delforge M, Kobbe G, Selleslag D, Schouten HC, Ferrant A, Biersack H, Amadori S, Muus P, Jansen JH, Hellstrom-Lindberg E, Kovacsovics T, Wijermans P, Ossenkoppele G, Gratwohl A, Marie JP, Willemze R. Value of allogeneic versus autologous stem cell transplantation and chemotherapy in patients with myelodysplastic syndromes and secondary acute myeloid leukemia. Final results of a prospective randomized European Intergroup Trial. Haematologica. 2010 Oct;95(10):1754-61. doi: 10.3324/haematol.2009.019182. Epub 2010 May 21. PMID 20494931